CLINICAL TRIAL: NCT06534606
Title: Additional Effects of Sternocleidomastoid Release With SNAGS in the Management of Cervicogenic Headache
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/17
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Cervicogenic Headache
MeSH Terms: conditions — Post-Traumatic Headache | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial having two groups. One group will receive SNAGs and the second will receive Sternocleidomastoid Release along with SNAGS. Both groups will be recruited concurrently.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional physical therapy Group (Active Comparator): Both Group A and Group B will receive this conventional physical therapy protocol for cervicogenic headache.
  * Moist heat therapy: Frequency: 15 minutes, 3 times per week (alternatively) for 2 weeks.
  * TENS application: Frequency: 15 minutes, 3 times per week (alternatively) for 2 weeks.
  In addition to this, they will receive Headache SNAGs (Sustained Natural Apophyseal Glides) 5 sets of 10 repetitions. Each repetition will be given with a 10 second hold.
  • Frequency: 3 times a week for 2 weeks. 6 sessions in total.
  Interventions: Procedure: Electrotherapy and physical agents; Procedure: Headache SNAGs
- Conventional physical therapy with sternocleidomastoid release (Experimental): Both Group A and Group B will receive this conventional physical therapy protocol for cervicogenic headache.
  * Moist heat therapy: Frequency: 15 minutes, 3 times per week (alternatively) for 2 weeks.
  * TENS application: Frequency: 15 minutes, 3 times per week (alternatively) for 2 weeks.
  Headache SNAGs: In addition to the conventional physical therapy protocol, they will receive Headache SNAGs (Sustained Natural Apophyseal Glides) 5 sets of 10 repetitions. Each repetition will be given with a 10 second hold.
  * Frequency: 3 times a week for 2 weeks. 6 sessions in total. Sternocleidomastoid Release: Group B will also receive Sternocleidomastoid release in addition with headache SNAGs. Release to the sternocleidomastoid muscle will be given once per session for 5-8 minutes.
  * Frequency: 3 times a week for 2 weeks. 6 sessions in total.
  Interventions: Procedure: Electrotherapy and physical agents; Procedure: Headache SNAGs; Procedure: Sternocleidomastoid Release

INTERVENTIONS:
Procedure: Electrotherapy and physical agents — Moist heat therapy: Frequency: 15 minutes, 3 times per week (alternatively) for 2 weeks.
  • TENS application: Frequency: 15 minutes, 3 times per week (alternatively) for 2 weeks.
Procedure: Headache SNAGs — Headache SNAGs (Sustained Natural Apophyseal Glides) 5 sets of 10 repetitions. Each repetition will be given with a 10 second hold.
  • Frequency: 3 times a week for 2 weeks. 6 sessions in total.
Procedure: Sternocleidomastoid Release — Sternocleidomastoid Release: Group B will also receive Sternocleidomastoid release in addition with headache SNAGs. Release to the sternocleidomastoid muscle will be given once per session for 5-8 minutes.Frequency: 3 times a week for 2 weeks. 6 sessions in total.
  Arms: Conventional physical therapy with sternocleidomastoid release

SUMMARY:
Cervicogenic headache is a common type of headache in adults which causes disability and difficulty in everyday activities. According to the latest International Headache Society model, cervicogenic headache (CGH) is a secondary headache having C1-C2 dysfunction. SNAGs are highly effective in the treatment approach for these patients. Sternocleidomastoid muscle receive overactive tension from forward neck posture, increasing muscular fatigue and tone of muscles. This tension in SCM causes referred pain in the head and neck region. SNAGs are very effective but musculoskeletal impairments especially the tightness of sternocleidomastoid muscle still persist and can exacerbate symptoms. Manual therapy targeted to the SCM muscle may be effective for reducing headache and neck pain intensity and increasing performance of deep cervical flexors. Findings of this study will aid the therapists in choosing which technique to use while treating the patients. This will save therapist's time and effort as they will not be using the less effective treatment protocol. Furthermore, patient's time and investment will be used in the right direction.

ELIGIBILITY:
Inclusion Criteria:

* Age group: 18-45 years old
* Both males and females
* Unilateral headache with no shift of side
* C1-C2 Dysfunction
* Positive flexion rotation test (Rotation restriction is greater than 10 degrees)
* Headache at least once a month in the last 3 months
* Headache with at least 4 score in NPRS (Sign and Symptoms of Neck Involvement)
* Headache with restriction of ROM in the neck
* Headache precipitated by:

Sustained neck movements, and awkward head positioning. External Pressure over upper cervical or occipital region

Headache Characteristics:

* Moderate-severe, non-throbbing pain, usually starting in the neck.
* Episodes of varying duration, or: fluctuating, continuous pain

Exclusion Criteria:

* Headache of non-cervical origin
* Diagnosed Cases of:Cervical spondylosis,Cervical radiculopathy/ nerve root involvement/ disc herniation,Cervical instability/ fracture,Vertebrobasilar insufficiency ,Cervical spine surgery,Cervical spondylolisthesis,Spinal infection or tumors,Osteoporosis,History of trauma,Rheumatoid Arthritis,Inflammatory Arthritis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 2 weeks
  Pain will be measured on the basis of Numeric Pain Rating Scale score.
Range of motion | 2 weeks
  Cervical rotation will be measured through CROM device
Headache Disability | 2 weeks
  Headache Disability Index will be used
Cervical Proprioception | 2 weeks
  Joint Position Error Test will be used

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan